CLINICAL TRIAL: NCT04669912
Title: Observational Study of Glycemic Control and Self-management of Young People (Aged 13 to 25 Years ) With Type 1 Diabetes During COVID-19 Lockdown.
Brief Title: COVID-19 Pandemic Lockdown Effect in Adolescents and Young Adults With Type 1 Diabetes: Positive Results of an Unpreceded Challenge for Telemedicine and Patient Self-management
Acronym: COVIDIABADO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: IDRCB 2020-A02760-39
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; adolescent; COVID-19; telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: glucose control and sensor usage — Data related to glucose control and sensor usage collected from the Libreview platform

SUMMARY:
Lockdown resulting from the COVID-19 pandemic was an unpreceded model of the impact of lifestyle on chronic diseases, especially for adolescents and young adults with type 1 diabetes (T1D) whose lifestyle is known to strongly impact disease management. The investigators aimed to assess changes in self-monitoring and glycemic control in this population before, during, and after the two-month French lockdown. Te investigators hypothesized an improvement in glucose control and glucose sensor usage.

The protocol will include all patients with T1D from 13 to 25 years old using a flash glucose monitoring related to the LibreView cloud platform.

The primary outcome, evolution of percentage of glucose time in range 70-180 mg/dL (TIR), and secondary outcomes (glucose management indicator GMI, time spent below range TBR, and sensor usage) will be analyzed with a linear mixed-effects regression model.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) data will be collected from the cloud-based platform, LibreView.

Data will be collected for patients from Sud-Francilien hospital (Corbeil-Essonnes, France) and Kremlin-Bicêtre hospital (Kremlin-Bicêtre, France). Data related to glucose control and sensor usage will be collected from the Libreview platform. Data related to patients' characteristics, treatment and telemedicine visits (number of contacts with health professionals) will be collected from the medical record and confirmed with telephone-administered questionnaire.

The lockdown imposed by the French government occurred from March 17 to May 10, 2020. Therefore, outcomes will be assessed 4 times: the month before lockdown, during the first month, the second month of lockdown, and one month after lockdown ended.

Potential confounding factors will be studied: age, gender, type of insulin delivery (multiple daily injections, MDI; insulin pump), contacts with health professionals (physician or nurse).

Descriptive statistics will include means with standard deviations, numbers of patients and percentages.

Outcomes will be analysed with a linear mixed-effects regression model. Analyses will be performed with R studio version 3.5.0.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age between 13 and 25 years
* use of a flash glucose monitoring related to the LibreView cloud platform
* patients follow-up by the diabetes department of Hopital Sud Francilien or the diabetes department of Hôpital Bicêtre.
* patient informed of the study and not having objected to it.

Exclusion Criteria:

* patients out of France during lockdown
* other type of diabetes
* Duration of diabetes of less than one year
* patient aged under 13 years or above 26 years old

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population will be selected from two university general hospitals of the region of Ile de France (France): Kremlin-Bicetre hospital and Sud-Francilien hospital.
  The population will be aged from to 13 to 25 years at the beginning of lockdown.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Changes in percentage of time spent in range 70-180 mg/dL after lockdown compared to before lockdown | Measure repeated 2 times : month before lockdown (28 days), after lockdown
  Percentage of time spent in glucose range from 70 to 180 mg/dL over a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Changes in percentage of time spent in range 70-180 mg/dL during first month of lockdown compared to before lockdown | Measure repeated 2 times : month before lockdown (28 days), first month of lockdown (28 days)
  Percentage of time spent in glucose range from 70 to 180 mg/dL over a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Changes in percentage of time spent in range 70-180 mg/dL during second month of lockdown compared to before lockdown | Measure repeated 2 times : month before lockdown (28 days), second month of lockdown (28 days)
  Percentage of time spent in glucose range from 70 to 180 mg/dL over a month (28 days) according to continuous glucose monitoring data collected on Libreview.

SECONDARY OUTCOMES:
Evolution of glucose management indicator (GMI) compared to before lockdown. | Measures repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Glucose Management Indicator (GMI) approximates the laboratory A1C level expected based on average glucose measured using continuous glucose monitoring data collected on Libreview.
Evolution of glucose time spent below range <54 mg/dL | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Percentage of time spent in this glucose range in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of glucose time spent below range 54 - 70 mg/dL | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Percentage of time spent in this glucose range in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of glucose time spent below range 180-250 mg/dL | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Percentage of time spent in this glucose range in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of glucose time spent below range > 250 mg/dL | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Percentage of time spent in this glucose range in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of average glucose in mg/dL compared to before lockdown. | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Average glucose level in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of hypoglycaemia frequency compared to before lockdown. | Measure repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  Number of hypoglycaemia events (glycemia under 70 mg/dL during at least 15 minutes) in a month (28 days) according to continuous glucose monitoring data collected on Libreview.
Evolution of glucose sensor use compared to before lockdown. | Measures repeated 4 times (including 28 days of data for each): month before lockdown (28 days), first month of lockdown (28 days), second month of lockdown (28 days), first month after lockdown (28 days).
  The level of glucose data collected related to the glucose monitoring frequency and the number of scans with continuous glucose monitoring data collected on Libreview.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred PENFORNIS, MD PhD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No